CLINICAL TRIAL: NCT06513637
Title: 12-Lead ECG Database
Brief Title: 12 Lead ECG Database
Status: Not yet recruiting | Type: Observational
Sponsor: Huxley Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-10002 12 Lead ECG Database
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: 12-Lead ECG and home sleep study (HST) diagnostics — * 12-lead ECG hookup will be performed following standard placement procedures.
  * The Home Sleep Study diagnostic device placement will be performed by study personnel following the manufacturer's instructions.

SUMMARY:
The purpose of this investigation is to collect a database of simultaneous electrocardiogram (ECG) recordings from the SANSA device and a reference 12-lead ECG recording device.

The purpose of this database is to aid development and evaluation of algorithms to detect cardiac arrhythmias and other parameters from the electrocardiogram. Example analyses that may utilize this database are ECG vector transformations and ECG waveform timing analyses.

The study is for scientific purposes and does not intend to diagnose, cure, mitigate, treat, or prevent any disease and does not involve any medical procedures.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older.
* are able to read, understand, and sign informed consent documentation.
* are willing to undergo simultaneous recordings with the Sansa and 12-lead ECG device.

Exclusion Criteria:

* exhibit deformities of the chest (e.g., pronounced scarring, pectus carinatum) that would interfere with sensor placement
* have broken or injured skin that would interfere with sensor placement
* are known to experience adverse reactions to medical-grade adhesive
* are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will receive the same treatment; there are no groups or cohorts that receive different treatments. Study populations at each site will be enrolled from patients, site personnel, or the general population. Recruitment may, from time to time, target enrichment of a particular demographic, subject characteristic, or cardiac arrhythmia to increase the diversity and representation of the database.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-19 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
No specified primary endpoint | Subjects will participate in a single visit. Subjects will be considered enrolled upon signing the informed consent. The entire duration of enrollment is expected to be less than one hour and no more than six hours
  This data collection protocol does not have any specific data analysis endpoints. Its purpose is to collect data to be included in an ECG database that may be used for various future analyses.
  The number, severity, and device/comparator relatedness of AEs reported while subjects undergo study procedures will be reported.

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared to other researchers.